CLINICAL TRIAL: NCT02998853
Title: Reliability of 3D Angio QFR Evaluation of Non Culprit Stenoses in STEMI Patients During First Acute Interventional Procedure: Comparison With Staged Procedure FFR
Brief Title: Non Culprit Functional Evaluation With 3D Angio QFR in STEMI PCI Procedure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Sant'Anna e San Sebastiano (Other)
Responsible Party: Principal Investigator, dr. Domenico Di Girolamo, MD, Azienda Ospedaliera Sant'Anna e San Sebastiano
Other Study IDs: AOStAnnaSS
Record Dates: First submitted 2016-12-13; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Percutaneous Coronary Intervention; Coronary Artery Disease
Keywords: Non culprit; STEMI PCI; angio QFR; FFR; Staged procedure
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: QFR measurement by dedicated workstation on xrays angio selected runs — The patient undergoes coronary angiography; if at least one stenosis from 40 to 90% in non culprit is present and FFR is indicated by guidelines the patient is enrolled to 3d Angio QFR evaluation; no adjunctive invasive procedures are needed for QFR measurements
  Other Names: 3d Angio QFR evaluation

SUMMARY:
Reliability of 3D angio QFR functional evaluation of all non culprit lesions >50% in STEMI patients during first acute procedure

DETAILED DESCRIPTION:
3DAngio QFR is an angiographic based tool for coronary stenosis functional assessment: it is validated versus Adenosine FFR(ADOFFR) by several studies (FAVOR, VIRTU-1) ; in particular post contrast QFR (cQFR) showed a very good correlation with ADOFFR. Furthermore ADOFFR in non culprit vessel in acute stage of STEMI correlates well with ADOFFR of the same non culprit lesion in staged procedure. Aim of the study is to find a valid correlation between cQFR in acute study and ADOFFR in the staged procedure. A positive result may lead to a fast, easy and cost effective acute functional non culprit lesions evaluation during acute procedure for STEMI patients, selecting those,if any, to be treated immediately or in a staged procedure.

ELIGIBILITY:
Inclusion Criteria:

* STEMI/NSTEMI pts with at least 1 non culprit lesion > 50%
* Age > 18 years
* Able to provide signed informed consent
* Angiographic inclusion criteria:
* Indication for FFR in at least one stenosis:
* Diameter stenosis of 50%-90% by visual estimate
* Reference vessel size > 2 mm in stenotic segment by visual estimate

Exclusion Criteria:

* Severe asthma or severe chronic obstructive pulmonary disease
* Severe heart failure (NYHA≥III)
* S-creatinine>150µmol/L or GFR<45 ml/kg/1.73m2
* Allergy to contrast media or adenosine
* Atrial fibrillation

Angiographic exclusion criteria:

poor coronary opacification marked overlapping marked tortuosity angio acquisition protocol incomplete

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive STEMI patients with at least one non culprit artery with stenosis >50%.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of TIMI flow based with contrast hyperemia QFR in acute study comparison to FFR in staged procedure reported as positive and negative likelihood ratio in the same lesion | 1 - 15 days
  Diagnostic performance of QFR in comparison to FFR reported as positive and negative likelihood ratio

SECONDARY OUTCOMES:
Diagnostic accuracy of TIMI flow based for computing QFR in acute study in comparison with TIMI flow based for computing QFR in staged in the same lesion | 0-15 days
  Diagnostic accuracy of TIMI flow based for computing QFR in acute study in comparison with TIMI flow based for computing QFR in staged in the same lesion
Diagnostic accuracy of TIMI flow based for computing QFR in staged study in comparison with Hyperemic FFR in the same lesion | 0-1 hour
  Diagnostic accuracy of TIMI flow based for computing QFR in acute study in comparison with TIMI flow based for computing QFR in staged in the same lesion

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Di Girolamo, Principal Investigator — Azienda Ospedaliera Sant'Anna e San Sebastiano; Giuseppe MERCONE, MD, Principal Investigator — Azienda Ospedaliera Sant'Anna e San Sebastiano
Locations (1):
- Azienda Ospedaliera Sant-Anna e San Sebastiano, Caserta, Caserta, Italy

REFERENCES:
- [Result] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Result] Safi M, Eslami V, Namazi MH, Vakili H, Saadat H, Alipourparsa S, Adibi A, Movahed MR. Visual-Functional Mismatch Between Coronary Angiography, Fractional Flow Reserve, and Quantitative Coronary Angiography. Int J Angiol. 2016 Dec;25(4):229-234. doi: 10.1055/s-0035-1569992. Epub 2015 Dec 31. PMID 27867288
- [Result] Gaur S, Taylor CA, Jensen JM, Botker HE, Christiansen EH, Kaltoft AK, Holm NR, Leipsic J, Zarins CK, Achenbach S, Khem S, Wilk A, Bezerra HG, Lassen JF, Norgaard BL. FFR Derived From Coronary CT Angiography in Nonculprit Lesions of Patients With Recent STEMI. JACC Cardiovasc Imaging. 2017 Apr;10(4):424-433. doi: 10.1016/j.jcmg.2016.05.019. Epub 2016 Oct 12. PMID 27743953
- [Result] Indolfi C, Mongiardo A, Spaccarotella C, Torella D, Caiazzo G, Polimeni A, Sorrentino S, Micieli M, Sabatino J, Curcio A, De Rosa S. The instantaneous wave-free ratio (iFR) for evaluation of non-culprit lesions in patients with acute coronary syndrome and multivessel disease. Int J Cardiol. 2015 Jan 15;178:46-54. doi: 10.1016/j.ijcard.2014.03.210. Epub 2014 Oct 28. PMID 25464218
- [Result] Sulimov DS, Abdel-Wahab M, Richardt G. Fractional Flow Reserve in Acute Myocardial Infarction: A Guide for Non-Culprit Lesions? Cardiol Ther. 2015 Jun;4(1):39-46. doi: 10.1007/s40119-015-0040-4. Epub 2015 Jun 9. PMID 26055262
- [Result] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Result] Morris PD, Ryan D, Morton AC, Lycett R, Lawford PV, Hose DR, Gunn JP. Virtual fractional flow reserve from coronary angiography: modeling the significance of coronary lesions: results from the VIRTU-1 (VIRTUal Fractional Flow Reserve From Coronary Angiography) study. JACC Cardiovasc Interv. 2013 Feb;6(2):149-57. doi: 10.1016/j.jcin.2012.08.024. PMID 23428006
- [Result] Morris PD, van de Vosse FN, Lawford PV, Hose DR, Gunn JP. "Virtual" (Computed) Fractional Flow Reserve: Current Challenges and Limitations. JACC Cardiovasc Interv. 2015 Jul;8(8):1009-1017. doi: 10.1016/j.jcin.2015.04.006. Epub 2015 Jun 24. PMID 26117471
- [Result] Papafaklis MI, Muramatsu T, Ishibashi Y, Lakkas LS, Nakatani S, Bourantas CV, Ligthart J, Onuma Y, Echavarria-Pinto M, Tsirka G, Kotsia A, Nikas DN, Mogabgab O, van Geuns RJ, Naka KK, Fotiadis DI, Brilakis ES, Garcia-Garcia HM, Escaned J, Zijlstra F, Michalis LK, Serruys PW. Fast virtual functional assessment of intermediate coronary lesions using routine angiographic data and blood flow simulation in humans: comparison with pressure wire - fractional flow reserve. EuroIntervention. 2014 Sep;10(5):574-83. doi: 10.4244/EIJY14M07_01. PMID 24988003